CLINICAL TRIAL: NCT04920396
Title: Intense Regulated Pulsed Light Vs Standard of Care for the Treatment of Meibomian Gland Dysfunction
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-Investigator not available
Sponsor: Aston University (Other)
Responsible Party: Principal Investigator, James Wolffsohn, Professor, Aston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eeye03182021
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized allocation between treatments
Who Masked: Investigator
Masking Description: Ocular assessment will be undertaken by a researcher masked to the participants treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IRPL (Experimental): Three treatments with IRPL (manufacturer: E-Swin, France) on days 0, 15 and 45
  Interventions: Device: E>Eye IRPL
- Warm compress (Active Comparator): Daily use of a warm compress (manufacturer: The Eye Doctor, UK) with Sterileyes® twice a day for 5 minutes
  Interventions: Device: Warm compress

INTERVENTIONS:
Device: E>Eye IRPL — Regulated intense pulsed light therapy
  Arms: IRPL
Device: Warm compress — Fabric mask with anti-bacterial coating filled with BodyBeads® heated in a microwave for 30 seconds before application over the eyes for 5 minutes
  Other Names: The Eye Doctor Mask
  Arms: Warm compress

SUMMARY:
This study is to evaluate the effectiveness of E>EYE intense regulated pulsed light (IRPL) treatment compared to the current standard of care using a daily warm compress

DETAILED DESCRIPTION:
E-Eye is a medical device that has been specifically designed for treating dry eye syndrome due to meibomian gland dysfunction (MGD). This study is a prospective, single centred, interventional, randomized study assessing the efficacy and safety of E>EYE in the management of MGD (3 applications on days 0, 15 and 45, with a follow up 1 month later) compared to daily use of a warm compress over a period of 75 days.

The study will monitor the change in symptoms and signs of dry eye at each visit.)

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and participate in the required study visit
* Subjects determined to have signs and symptoms of evaporative Dry Eye disease due to MGD, defined by the following:

  * OSDI score >13 and
  * NITBUT <= 10sec

Exclusion Criteria:

* No use of warm compresses, intense pulsed light therapy or other lid warming treatment in the past 6 Months
* Patients with greater 75% meibomian gland loss
* Presence of ocular pathology or systemic conditions other than previously diagnosed moderate or severe chronic dry eye and/or Sjogren's syndrome, that in the investigator's judgment may affect the testing for, or diagnosis of, dry eye if present
* Use of prescribed ocular topical medication (e.g., anti-hypertensive, steroid, Cyclosporin A, antibiotic) within the last 24 hours
* Artificial tear usage within 2 hours prior to study testing
* Other invasive ocular diagnostic testing within 2 hours prior to study testing
* Eye makeup present on the eye lid within 10 minutes prior to study testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Symptoms of dry eye disease | Change between baseline and day 75
  Change in Ocular Surface Disease Index (OSDI) questionnaire score from baseline to end of trial
Tear film stability | Change between baseline and day 75
  Change in non-invasive assessed tear film retention time from baseline to end of trial

SECONDARY OUTCOMES:
Eye redness | Change between baseline and day 75
  Change in ocular redness graded against standardised Efron grading scale (from 0 to 4, where lower is better)
Meibomian gland patency | Change between baseline and day 75
  Change in the number of glands expressing multiplied by the quality (on a 4 point standardised scale)
Tear volume | Change between baseline and day 75
  Change in tear meniscus height measured in millimeters
Lipid layer thickness | Change between baseline and day 75
  Change in white light interferometry pattern graded against the Guillon standardised categories (Open meshwork, closed meshwork, wave pattern, amorphous or colored fringes)

CONTACTS AND LOCATIONS:
Overall Officials: James Wolffsohn, PhD, Principal Investigator — Aston University
Locations (1):
- Market Mall Eye Clinic - Calgary, AB, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No